CLINICAL TRIAL: NCT07052916
Title: Pilot Trial of Telehealth Music Therapy for Cognitive Dysfunction in Hematologic Cancer Survivors (PRELUDE)
Brief Title: A Music Therapy Study for Blood Cancer Survivors With Cognitive Difficulties
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-119
Record Dates: First submitted 2025-06-30; First posted 2025-07-08 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Blood Cancer; Lymphoma; Leukemia; Myeloma
Keywords: Blood cancer survivor; myeloma; Leukemia; Lymphoma; Memorial Sloan Kettering Cancer Center; 25-119
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma; Leukemia; Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music Therapy/MT (Experimental): Participants will receive 12, weekly 60-minute MT sessions (+/- 1 week) with homework in-between sessions to reinforce in-session concepts, practice musical skills, and serve as transitions to subsequent sessions
  Interventions: Other: Music Therapy/MT
- Therapist Attention-Music Education/TAME control (Active Comparator): Patients will receive 12, weekly 60-minute Therapist Attention-Music Education/TAME sessions (+/- 1 week) with homework in-between sessions to reinforce in-session concepts and serve as transitions to subsequent sessions. The TAME control group will involve board-certified music therapists guiding participants through music listening exercises.
  Interventions: Other: Therapist-Attention Music Education/TAME Control
- Wait-List Control/WLC (No Intervention): The Wait-List Control/WLC group will receive usual care from healthcare providers and complete the same assessments as the other groups. The WLC will have the option of receiving either 12 sessions of MT or 12 sessions of TAME intervention when the study concludes after the 24-week waiting period. The WLC participants will choose which intervention (MT or TAME) they wish to receive.

INTERVENTIONS:
Other: Music Therapy/MT — Therapeutic music lessons are the core component of the Music Therapy/MT intervention. Other components include guided music listening to help participants use music as a tool for regulating mood, energy, and attention, as well as music-centered discussions to help participants discover songs with personal meaning that they will enjoy learning to play.
  Arms: Music Therapy/MT
Other: Therapist-Attention Music Education/TAME Control — Participants will receive 12, weekly 60-minute TAME sessions (+/- 1 week) with homework in-between sessions to reinforce in-session concepts and serve as transitions to subsequent sessions. The TAME control group will involve board-certified music therapists guiding participants through music listening exercises.
  Arms: Therapist Attention-Music Education/TAME control

SUMMARY:
Research has shown that music-based activities may help improve brain functions, such as attention, memory, and executive function. Because of this past research, the researchers are doing this study to find out whether telehealth music therapy is a practical treatment for cognitive difficulties in blood cancer survivors. The researchers will also study whether music therapy and music education help improve cognitive function and other common symptoms such as anxiety, depression, and/or tiredness.

ELIGIBILITY:
Inclusion Criteria:

* English-proficient, aged 18 or older
* Diagnosis of lymphoma, leukemia, or myeloma
* Stable oncologic disease or no evidence of disease as indicated in the medical chart or by the oncology team
* Score of <54 on the FACT-Cog PCI subscale
* Minimum life expectancy of one year as per clinician assessment
* Patient should be able to understand and complete all study assessments on their own.
* Eligible patient should be able to understand informed consent and provide signed informed consent in English.

Exclusion Criteria:

* Less than 3 months since completion of surgery, radiation, induction chemotherapy (for newly diagnosed or relapsed disease), transplantation, or immunotherapy (e.g., CAR T-Cell, bispecific antibodies)

  * If there is a defined treatment period, the patient must be at least 3 months from treatment completion
  * If the patient is on continuous therapy, patient must have completed at least 6 months of the therapy
  * Maintenance therapies are allowed
* Received music therapy (MT) in the past year
* Current music training, >6 months of music training in the past 10 years, or plan to initiate music training during the study
* No access to an internet-connected device
* Active suicidal ideation, bipolar, schizophrenia, or substance abuse
* BOMC score ≥10 (indicative of dementia)
* Uncorrectable visual, auditory, or motor impairments
* Initiation or altered dose of sedative, stimulant, or anti-cholinergic medications in the past month or plan to initiate these medications during the study, as these are known to impact cognitive function
* Initiation of any other interventions for CRCD (e.g., cognitive rehabilitation) in the past month or plan to initiate these interventions during the study, as these are known to impact cognitive function

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-12-27 (Estimated); Study Completion 2026-12-27 (Estimated)

PRIMARY OUTCOMES:
Feasibility of studying a telehealth-based Music Therapy/MT intervention for cancer-related cognitive dysfunction/CRCD in hematologic cancer survivors as defined as the completion of 9 or more sessions. | up to 1 year
  The primary objective of this study is to determine the feasibility of studying a telehealth-based Music Therapy/MT intervention for cancer-related cognitive dysfunction/CRCD in hematologic cancer survivors. Feasibility will be defined as the completion of 9 or more sessions out of the planned 12 weekly sessions of music therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Liou, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All protocol activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All protocol activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center Suffolk - Commack (All protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All protocol activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All protocol activities), New York, New York
  - Memorial Sloan Kettering Nassau (All protocol activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org